CLINICAL TRIAL: NCT02759055
Title: Improving Prediabetes Cardiovascular Care With EHR-Based Decision Support
Brief Title: Pre-Diabetes Cardiovascular (CV) Care (Pre-Diabetes Wizard)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: Essentia Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HL128614-01
Record Dates: First submitted 2016-04-27; First posted 2016-05-03 (Estimated); Results first posted 2021-03-16 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2020-12

CONDITIONS: Pre-diabetes
MeSH Terms: conditions — Glucose Intolerance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clinical Decision Support (CV Wizard) (Experimental): In the Intervention arm, primary care providers will be provided with an EHR-linked, Web-based clinical decision support system that identifies patients with prediabetes and provides patients and their primary care providers personalized, evidence-based CDS and follow up to reduce risk of heart attacks or stroke, optimizing management and follow up of pre-diabetes patients with uncontrolled CV risk factors.
  Interventions: Other: Clinical Decision Support
- Usual Care (No Intervention): In the No Intervention arm, patients receive usual care from their primary care clinic and care providers.

INTERVENTIONS:
Other: Clinical Decision Support — an EHR-linked, Web-based clinical decision support (CDS) system that identifies patients with prediabetes and provides patients and their primary care providers personalized, evidence-based CDS and follow up to reduce risk of heart attacks or stroke
  Other Names: CV Wizard
  Arms: Clinical Decision Support (CV Wizard)

SUMMARY:
Nearly one in three adults has prediabetes, a condition that substantially increases the risk of heart attacks and stroke. The increased cardiovascular risk associated with prediabetes can be effectively managed by lifestyle changes or medication therapy, but recent data shows few prediabetes patients are treated effectively. In this project, we will adapt, implement, and evaluate a proven electronic health record-linked, web-based clinical decision support system to identify patients with prediabetes and provide prioritized treatment recommendations to patients and providers in a rural health system. The results of the project will provide a template for implementation of more efficient and effective rural healthcare and have the potential to substantially and improve cardiovascular quality of care and clinical outcomes of millions of rural Americans with prediabetes.

DETAILED DESCRIPTION:
Nearly one in three adults in rural communities has prediabetes, a condition that increases the risk of heart attacks and stroke but can be managed by use of metformin, lifestyle interventions, and control of major cardiovascular (CV) risk factors. However, current prediabetes care is characterized by: (a) delayed recognition of prediabetes; (b) patient unawareness of effective treatment options for prediabetes; (c) poor control of concomitant major CV risk factors; (d) very low rates of metformin initiation; and (e) low rates of follow up to assess ongoing effectiveness of prediabetes management.1-3 Increased use of electronic health records (EHR) in rural communities now provides a new opportunity to improve awareness and management of prediabetes and to reduce these patients' significant CV risk burden. In this project, we implement and evaluate an EHR-linked, Web-based clinical decision support (CDS) system that identifies patients with prediabetes and provides patients and their primary care providers personalized, evidence-based CDS and follow up to reduce risk of heart attacks or stroke. To accomplish this objective, we randomly allocate 30 primary care clinics with their 450 primary care providers and estimated 17,000 prediabetes patients to one of two intervention arms: Usual Care; or else the prediabetes CDS to optimize management and follow up of prediabetes patients with uncontrolled CV risk factors. Random-effects models assess intervention impact on: (a) American College of Cardiology/American Heart Association (ACC/AHA) pooled CV risk; (b) major CV risk factors (blood pressure, lipids, HbA1c, smoking, and BMI); (c) use of evidence-based drugs, including metformin, and lifestyle interventions to manage prediabetes; and (d) patient and provider satisfaction with the intervention strategy. We also conduct a state-of-the-art cost and a cost-effectiveness analysis of the interventions relative to usual care. The Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) framework, supplemented by the Consolidated Framework for Implementation Research (CFIR), is used to assess implementation processes and outcomes in a rural/urban health system.

The results of the project will provide a template for implementation of personalized CDS tools in rural and urban health settings, resulting in more efficient and effective rural healthcare that can be broadly applied across many clinical domains, incorporates patient treatment preferences, and has the potential to substantially improve the quality of CV care and clinical outcomes of millions of Americans with prediabetes residing in medically underserved areas.

ELIGIBILITY:
Inclusion Criteria:

* Pre-Diabetes Diagnosis or Clinical Lab Values and
* One or more of the following CV risk factors: Current smoking, Hypertension, elevated LDL, or BMI not within normal range, AND
* at least one subsequent primary care visit to a randomized clinic 12 to 24 months after the index visit.

Exclusion Criteria:

* Evidence of Diabetes in the previous 12 months
* Pregnant
* Hospice care or Chemotherapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21664 (Actual)
Dates: Start 2016-10; Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Saman, PhD, Principal Investigator — Essentia Institute of Rural Health
Locations (1):
- Essentia Health, Duluth, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Karve A, Hayward RA. Prevalence, diagnosis, and treatment of impaired fasting glucose and impaired glucose tolerance in nondiabetic U.S. adults. Diabetes Care. 2010 Nov;33(11):2355-9. doi: 10.2337/dc09-1957. Epub 2010 Aug 19. PMID 20724649
- [Derived] Saman DM, Allen CI, Freitag LA, Harry ML, Sperl-Hillen JM, Ziegenfuss JY, Haapala JL, Crain AL, Desai JR, Ohnsorg KA, O'Connor PJ. Clinician perceptions of a clinical decision support system to reduce cardiovascular risk among prediabetes patients in a predominantly rural healthcare system. BMC Med Inform Decis Mak. 2022 Nov 19;22(1):301. doi: 10.1186/s12911-022-02032-z. PMID 36402988
- [Derived] Pratt R, Saman DM, Allen C, Crabtree B, Ohnsorg K, Sperl-Hillen JM, Harry M, Henzler-Buckingham H, O'Connor PJ, Desai J. Assessing the implementation of a clinical decision support tool in primary care for diabetes prevention: a qualitative interview study using the Consolidated Framework for Implementation Science. BMC Med Inform Decis Mak. 2022 Jan 15;22(1):15. doi: 10.1186/s12911-021-01745-x. PMID 35033029

RESULTS

PARTICIPANT FLOW:
Groups:
- Clinical Decision Support (CV Wizard): In the Intervention arm, primary care providers will be provided with an Electronic Health Record-linked, Web-based clinical decision support system that identifies patients with prediabetes and provides patients and their primary care providers personalized, evidence-based CDS and follow up to reduce risk of heart attacks or stroke, optimizing management and follow up of pre-diabetes patients with uncontrolled cardiovascular risk factors.
  Clinical Decision Support: an Electronic Health Record(EHR)-linked, Web-based clinical decision support(CDS) system that identifies patients with prediabetes and provides patients and their primary care providers personalized, evidence-based CDS and follow up to reduce risk of heart attacks or stroke
Period: Overall Study
Arm/Group | Clinical Decision Support (CV Wizard) | Usual Care
Started | 12702 | 8962
Completed | 10775 | 7454
Not Completed | 1927 | 1508
Not completed — Patients with no follow-up visit and/or age 18-39 were not included in analyses. | 1927 | 1508

BASELINE CHARACTERISTICS:
Population: The population included in the analyses are those who had at least one follow-up visit and are age 40-75 at the time of the index visit.
Groups:
- Clinical Decision Support (Cardiovascular Wizard): In the Intervention arm, primary care providers will be provided with an Electronic Health Record-linked, Web-based clinical decision support system that identifies patients with prediabetes and provides patients and their primary care providers personalized, evidence-based Clinical Decision Support and follow up to reduce risk of heart attacks or stroke, optimizing management and follow up of pre-diabetes patients with uncontrolled cardiovascular risk factors.
  Clinical Decision Support: an Electronic Health Record-linked, Web-based clinical decision support (CDS) system that identifies patients with prediabetes and provides patients and their primary care providers personalized, evidence-based CDS and follow up to reduce risk of heart attacks or stroke
- Total: Total of all reporting groups
Arm/Group | Clinical Decision Support (Cardiovascular Wizard) | Usual Care | Total
Number analyzed (Participants) | 10775 | 7454 | 18229
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6331 | 4713 | 11044
  >=65 years | 4444 | 2741 | 7185
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (8.8) | 60.5 (8.8) | 60.9 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5428 | 3808 | 9236
  Male | 5347 | 3646 | 8993
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 49 | 30 | 79
  Not Hispanic or Latino | 10726 | 7424 | 18150
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 172 | 52 | 224
  Asian | 40 | 36 | 76
  Native Hawaiian or Other Pacific Islander | 7 | 2 | 9
  Black or African American | 77 | 38 | 115
  White | 10399 | 7299 | 17698
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 78 | 24 | 102
Region of Enrollment [Number; unit: participants]
  United States | 10775 | 7454 | 18229
Cardiovascular Risk [Mean (Standard Deviation); unit: units on a scale] — The American College of Cardiology/American Heart Association 10-year pooled atherosclerotic cardiovascular disease risk engine was used for 40-75 years olds, using the index visit values of systolic Blood Pressure, High Density Lipoproteins, total cholesterol, Body Mass Index, and smoking status. A lower result is better. Results range from Low-risk (<5%), Borderline risk (5% to 7.4%), Intermediate risk (7.5% to 19.9%), and High risk (≥20%). Statistical modeling to create the risk assessment tool was developed using a variety of participants from several large, diverse NHLBI-sponsored studies
  units on a scale | 11.2 (8.3) | 11.1 (8.4) | 11.2 (8.4)

OUTCOME MEASURES:

1. Primary Outcome: Predicted Annual Rate of Change in 10 Year Risk of Fatal or Nonfatal Heart Attack or Stroke
Description: 10-year cardiovascular risk was calculated at the index and all post-index patient encounters. A comparison of the difference in model-estimated annual rate of change in cardiovascular risk in Clinical Decision Support versus Usual Care clinics tested the primary efficacy hypothesis. The American College of Cardiology/American Heart Association (ACC/AHA) pooled CV risk calculator provides sex- and race-specific 10-year risk estimates for the first ASCVD event for black & white men & women aged 40-79 years. Variables included in risk assessment equations: age, total cholesterol, high-density lipoprotein cholesterol (HDL-C), systolic blood pressure (SBP) diabetes mellitus (diabetes), and current smoking status. 10-year risk for ASCVD categorized as: Low (<5%), Borderline (5% to 7.4%), Intermediate (7.5% to 19.9%), High (≥20%). Numerator: Rate of change in Clinical Decision Support. Denominator: Rate of change in Usual Care. Relative Risk < 1 supports primary hypothesis.
Time Frame: Index visit to 12 months post index visit
Population: The patients whose data were included in the primary outcome analysis were those who met eligibility criteria in the eligibility table.
Measure: Number (95% Confidence Interval); unit: units on a scale
Groups:
- Clinical Decision Support (CV Wizard): In the Intervention arm, primary care providers will be provided with an Electronic Health Record-linked, Web-based clinical decision support system that identifies patients with prediabetes and provides patients and their primary care providers personalized, evidence-based Clinical Decision Support and follow up to reduce risk of heart attacks or stroke, optimizing management and follow up of pre-diabetes patients with uncontrolled cardiovascular risk factors.
  Clinical Decision Support: an EHR-linked, Web-based clinical decision support (CDS) system that identifies patients with prediabetes and provides patients and their primary care providers personalized, evidence-based CDS and follow up to reduce risk of heart attacks or stroke
Arm/Group | Clinical Decision Support (CV Wizard) | Usual Care
Number analyzed (Participants) | 10775 | 7454
units on a scale | 1.100 [1.097 to 1.103] | 1.096 [1.029 to 1.101]
Statistical Analysis 1: Comparison: Clinical Decision Support (CV Wizard) vs Usual Care; Test type: Superiority; p < 0.05, Mixed Models Analysis; Risk Ratio (RR) = 1.003, 95% CI 2-sided [0.998 to 1.008]

ADVERSE EVENTS:
Time Frame: Up to 30 months
Groups:
- Clinical Decision Support (Cardiovascular Wizard): In the Intervention arm, primary care providers will be provided with an EHR-linked, Web-based clinical decision support system that identifies patients with prediabetes and provides patients and their primary care providers personalized, evidence-based CDS and follow up to reduce risk of heart attacks or stroke, optimizing management and follow up of pre-diabetes patients with uncontrolled cardiovascular risk factors.
  Clinical Decision Support: an EHR-linked, Web-based clinical decision support (CDS) system that identifies patients with prediabetes and provides patients and their primary care providers personalized, evidence-based CDS and follow up to reduce risk of heart attacks or stroke
Arm/Group | Clinical Decision Support (Cardiovascular Wizard) | Usual Care
All-Cause Mortality (participants affected / at risk) | 207/10775 | 159/7454
Serious Adverse Events (participants affected / at risk) | 1836/10775 | 1360/7454
Other Adverse Events (participants affected / at risk) | 339/10775 | 255/7454
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Clinical Decision Support (Cardiovascular Wizard) (N=10775) | Usual Care (N=7454)
Hospitalizations (General disorders) | 1836 | 1360 — It was pre-specified to monitor only hospitalizations and the laboratory values listed below for Serious and Other Adverse Events.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Clinical Decision Support (Cardiovascular Wizard) (N=10775) | Usual Care (N=7454)
Serum Potassium <= 3.0 mg/dl (Metabolism and nutrition disorders) | 138 | 97
Serum Potassium >= 6.5 mg/dl † (Metabolism and nutrition disorders) | 3 | 3
Serum Total CK >= 1200 mg/dl † (Musculoskeletal and connective tissue disorders) | 17 | 8
SBP < 90 mm Hg † (Vascular disorders) | 154 | 121
SBP >= 200 mm Hg † (Vascular disorders) | 40 | 36

LIMITATIONS AND CAVEATS:
CDS use was lower than the 80% target rate. Many patients had limited geographic or financial access to diabetes prevention programs. Due to differences in risk equations for patients age 40-75 (American College Cardiology/American Heart Association 10-year) and age 18-40 (Framingham 30 year), and missing lipid data in younger adults, the main analysis focused on age 40-75 years. Many with prediabetes had only modest potential for cardiovascular risk reductions clinicians may not prioritize.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-05): https://cdn.clinicaltrials.gov/large-docs/55/NCT02759055/Prot_SAP_000.pdf